CLINICAL TRIAL: NCT01300585
Title: MRI Evaluation to Assess the Relationship Between the Areolar Margin and Underlying Breast Paryenchyma Attachments to the Dermis
Brief Title: MRI Evaluation of the Breast Areolar Margin and Paryenchyma
Acronym: Breast MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Breast MRI
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Other): All patients on study will undergo an MRI of the breast(s).
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Patients who qualify for the study and consent to be included will undergo placement of areola and nipple markers that will be held in place with tape for the duration of the ordered MRI study. The markers consist of latex-free plastic tubing filled with vegetable based hydrogenated oil that is solid at room temperature. This creates a fat density marker that will define the areola but does not interfere with or create artifact onto the underlying tissue. The marker can be placed by the investigator or available MRI technician instructed in marker placement. The patient will then undergo the MRI. The patients participation in the study will end with the MRI.

SUMMARY:
The purpose of this study is to test a new method of defining patterns of how breast glands are or are not attached to the overlying skin. All patients will have markers placed on both breasts and will undergo an MRI. MRI results will be examined to identify the pattern of breast gland attachment to the overlying skin. This will help identify patients which may benefit from areolar sparing and/or nipple sparing technique and which patients should be treated by standard mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following indications for MRI study of the breast - screening for high risk without evidence of disease, have existing breast cancer with need for evaluation of extent of disease or to rule out additional occult cancer, or to have an equivocal mammogram or ultrasound requiring additional information from MRI.
* No prior breast surgery including prior excisional biopsies for disease performed with surgical technique, breast augmentation, reduction mammoplasty or breast lift with or without implants.
* Capable of fitting into the MRI machine.
* Permission to contact and consent the patient to participate from the investigator(s)
* Provide written informed consent and Authorization for Use/Disclosure of PHI

Exclusion Criteria:

* Have a contraindication to MRI study.
* Prior breast surgery - this includes: prior excisional biopsies for disease performed with surgical technique, breast augmentation, reduction mammoplasty or breast lift with or without implants [Patients may have undergone prior percutaneous (needle) biopsy or fine needle aspiration]
* Inability to fit into the MRI machine.
* Psychological factors that may interfere with successful completion of the study
* Refusal to provide written informed consent and/or Authorization for Use/Disclosure of PHI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Patterns of Breast Gland Attachment | 6 months
  Identify the various patterns of breast gland attachment to the overlying skin.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Richardson, MD, Principal Investigator — Piedmont Hospital
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States